CLINICAL TRIAL: NCT04774679
Title: Macroscopic on Cite Evaluation of EUS-FNA Specimen of Gastrointestinal Tumours With Everyday Needle (22g EUS FNA Needle)
Brief Title: Macroscopic on Cite Evaluation of EUS-FNA Specimen With 22 G Needle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hasan Yılmaz, Assistant Professor, Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MOSE
Record Dates: First submitted 2021-02-06; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: GI Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy Arm (Experimental): All patients who underwent EUS Guided biopsy
  Interventions: Procedure: Endosonographic fine needle aspiration biopsy

INTERVENTIONS:
Procedure: Endosonographic fine needle aspiration biopsy — An endoscopic ultrasound device will be inserted to the stomach and biopsy will performed with a needle

SUMMARY:
In order for the diagnosis of digestive system tumors and their appropriate treatment afterward, the type of these tumors should be determined by the pathologist. Pathology doctors need sufficient tissue (a small part of the organ thought to be diseased) to make a diagnosis. Tissue samples were taken from the patients by biopsy procedure. It is examined with microscopes by performing various staining and occasionally it is reported that sufficient tissue cannot be provided to make a diagnosis. In this case, patients may be subjected to repeated biopsy procedures. The aim of this study is to investigate whether the biopsy material obtained by endoscopic ultrasonography (EUS) is sufficient for the diagnosis of the pathology physician with the naked eye. Researchers will try to determine to what extent the physician performing the biopsy procedure can predict whether the tissue he has obtained is sufficient for the pathologist. In this way, researchers think that fewer biopsy repetitions will be needed in the future.

DETAILED DESCRIPTION:
This study was designed to improve the acquisition of sufficient tissue (EUS-FNA) with endosonography-assisted fine needle aspiration biopsy, which has been approved and used worldwide for the diagnosis of digestive system diseases. The procedure to be applied in the study is to determine the visible tissue fragments in the sample to be taken after the standard EUS-FNA procedure and to compare it with the diagnosis made by the pathologist. Patients with a tumor detected in the digestive system and referred to the investigation unit for tissue diagnosis will be included in this study. The data obtained in the study will be collected prospectively and will be analyzed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

1. İn the age range of 18-80 years old
2. Tumour detected withcross-sectional imagined technics in the digestive system

Exclusion Criteria:

1. Refuse to give written informed consent
2. Established bleeding disorder
3. INR>1.5IU plaelet count <100000/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of a macroscopically visible fragments in the 22g EUS-FNA needle specimens with final histologic diagnosis | 1-2 weeks
  Macroscopic appearance of the tissue fragments obtained by 22G EUS-FNA needle will be assessed by the endoscopist immediately in the endoscopy room. Endoscopits will decide the tissue acquisition is adequate. The diagnostic yield of the specimens determined by a pathologist will be compared to the endoscopist's first decision according to the macroscopic appearance.

SECONDARY OUTCOMES:
Area Under the size of the macroscopically visible core size versus histologic core size | 1-2 weeks
  Macroscopically visiable core size obtained via 22G EUS -FNA needle and pathologic size of cores will be compared by using

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at Mendeley data sharing platform freely and publicly
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 1 month after the study compilation
Access Criteria: publicly